CLINICAL TRIAL: NCT01517126
Title: Assessing Suicide Risk in Adolescents With Developmental Delays: Development of a Screening Tool
Brief Title: Assessing Suicide Risk in Adolescents With Developmental Delays
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912034; 12-M-N034
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Child Development Disorders, Pervasive
Keywords: Youth Suicide; Suicide Screening; Developmental Delay; Intellectual Disability; Assessment Instrument; Mental Retardation; Suicidal Thoughts; Suicidal Behavior
MeSH Terms: conditions — Child Development Disorders, Pervasive; Learning Disabilities; Intellectual Disability; Suicidal Ideation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

- Currently, there is no standard method to study suicide risk in youth with developmental delays or intellectual disabilities (DD/ID). Youth with DD/ID are often excluded from studies that are used to develop these methods. As a result, most current suicide risk assessments have not been tested for use with people with DD/ID. Researchers want to develop an effective suicide risk screening tool for children and adolescents with DD/ID.

Objectives:

- To develop a suicide risk screening tool for young adults with DD/ID.

Eligibility:

* Young adults between 12 and 21 years of age who have DD/ID and are in mental health counseling.
* Participants will be in counseling at Surrey Place Centre, a community health center in Toronto, Canada.

Design:

* Participants will fill out questionnaires during a 1-hour meeting with a therapist. The questions will ask about mood and current feelings, including whether the participant has been thinking about or planning to hurt or kill him or herself now or in the past. Other questions will ask about participants' understanding of death in general.
* Parents of participants may also fill out a questionnaire. It will ask about how the participant has been feeling. It will also ask whether the parent has noticed any signs that suggest suicidal thoughts or actions, now and in the past.
* Treatment will not be provided as part of this protocol. However, participants can receive counseling through the regular Surrey Place Centre services.

DETAILED DESCRIPTION:
Objective:

Currently, no gold standard is available for evaluating suicidal thoughts and behaviors in individuals with developmental delay or intellectual disabilities (DD/ID). Moreover, youth with DD are often excluded from instrument validation studies. Therefore, there is a paucity of sufficiently adapted and validated clinical suicide risk assessments for use with clients with DD/ID. The main objective of this study is to develop and assess the efficacy of a suicide screening tool for child and adolescent clients with DD/ID. More specifically:

Aim 1: To modify the Risk of Suicide Questionnaire (RSQ) in order to create a suicide screening tool for a pediatric mental health population with DD/ID.

Aim 2: To determine the feasibility of a suicide screening tool, (developed in Aim 1) to detect suicide risk in pediatric clients with DD/ID presenting to a community health center for mental health reasons.

Study population:

The NIMH is collaborating with Surrey Place Centre, a community health center in Toronto, Canada. The study population will be Surrey Place Centre clients, ages 12 and older, diagnosed with DD/ID, currently accessing individual mental health counseling. There will be no exclusion based on gender or race.

Design:

This will be a prospective instrument development study. Potential participants will be identified by research assistants (RAs) and therapists. Following informed consent and assent procedures, therapists will administer the Risk of Suicide Questionnaire Intellectual Disability Patient (RSQ-ID-Patient), and the Suicidal Ideation Questionnaire Child Version (SIQ-CV) to clients, and the RA will have the parents/guardians complete the Risk of Suicide Questionnaire-Intellectual Disability-Parent (RSQ-ID Parent). Three months after client participation, therapists will fill out a Therapist Follow-up Questionnaire.

Outcome measures:

Primary outcome measures include the RSQ-ID Patient, and the SIQ-CV, along with the RSQ-ID Parent. Secondary outcome measure is the Research Assistant Evaluation Form and the Clinician Follow- up Form.

ELIGIBILITY:
* INCLUSION CRITERIA:

Client must be enrolled in individual counseling at the Surrey Center at time of participation and must have attended at least 3 therapy appointments.

Clients must have an IQ score betwen 55 and 75 (a range considered to "mild developmental delay"). A client with mild DD will have the ability to communicate verbally and provide writtent assent. In order to receive services at Surrey Place Centre, clients must have a designation of "developmental delay" with and IQ score or range. If they do not have an IQ Score or DD designation, they undergo assessment at intake. Therefore, each client will have an IQ score recorded prior to study recruitment.

Age 12 years or older

English speaking

A legal guardian must provide informed consent and client must sign an assent document. Verbal assent is not acceptable for participation.

EXCLUSION CRITERIA:

Legal guradian is non-English speaking and no translation support is available to assist with the consent process.

No IQ score on record.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01-06; Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Horowitz, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- Surrey Place Centre, Toronto, Canada